CLINICAL TRIAL: NCT05635617
Title: Spatial Frequency Domain Imaging-based Perfusion Imaging to Assess Soft Tissue Injury in High Energy Lower Extremity Fracture
Brief Title: SFDI in High Energy Lower Extremity Fracture
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Dartmouth College (Other)
Responsible Party: Principal Investigator, Ida Leah Gitajn, Section Chief, Orthopaedics, Dartmouth-Hitchcock Medical Center
Other Study IDs: STUDY02001555
Record Dates: First submitted 2022-08-23; First posted 2022-12-02 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2024-07

CONDITIONS: Trauma Injury
Keywords: Trauma; Orthopaedic; Lower Extremity
MeSH Terms: conditions — Accidental Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Lower extremity fracture: High energy lower extremity fractures
  Interventions: Procedure: Lower Extremity Surgery

INTERVENTIONS:
Procedure: Lower Extremity Surgery — Patients 18 years of age or older with high energy lower extremity fractures. Provision of informed consent.

SUMMARY:
This is a non-randomized prospective study of 20 patients with high energy lower extremity fractures evaluating feasibility and acceptability of SFDI, a real-time optical imaging technology.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* High energy lower extremity fracture
* Provision of informed consent

Exclusion Criteria:

* Upper extremity fracture
* Metatarsal fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older who present to DHMC (Lebanon) with high energy lower leg trauma.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptability of the SFDI Imaging | 4 minutes or less
  The long-term objective for this research is to determine whether objective measures of perfusion through SFDI can be a predictive tool used in the ED, clinic or the operating room to determining when high-energy lower extremity fractures can safely undergo surgical fixation.

CONTACTS AND LOCATIONS:
Overall Officials: Ida L Gitajn, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No